CLINICAL TRIAL: NCT03872843
Title: A Prospective Double Blind Randomized Control Trial Comparing Opioid to Non-Opioid Protocol in Managing Postoperative Pain After Ureteroscopy With Stent Placement
Brief Title: Opioid Free Management After Ureteroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00056720
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Kidney Stone
Keywords: Ureteroscopy; Opioid; Non-Opioid; Stent Placement; Nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Analgesics, Opioid; Analgesics, Non-Narcotic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid Group (Active Comparator): This group includes subjects with renal stones who are consented for a ureteroscopy. They will be randomized to Norco 5milligram-325milligram Tablet for postoperative pain after ureteroscopy with stent placement.
  Interventions: Drug: Norco 5milligram-325milligram Tablet
- Non-Opioid Group (Active Comparator): This group includes subjects with renal stones who are consented for a ureteroscopy. They will be randomized to Ibuprofen 400 milligram for postoperative pain after ureteroscopy with stent placement.
  Interventions: Drug: Ibuprofen 400 MILLIGRAM in 1 TABLET ORAL TABLET, FILM COATED

INTERVENTIONS:
Drug: Norco 5milligram-325milligram Tablet — Designated coated 7 days supply of pain medication (Norco 5 milligram-325milligram Tablet) will be sent home with discharged subjects. Pain medication is administered/scheduled 4 times per day until the stent will be removed in clinic a week later.
  Other Names: Opioid
  Arms: Opioid Group
Drug: Ibuprofen 400 MILLIGRAM in 1 TABLET ORAL TABLET, FILM COATED — Designated coated 7 days supply of pain medication (Ibuprofen 400 milligram) will be sent home with discharged subjects. Pain medication is administered/scheduled 4 times a day as needed until the stent will be removed in clinic a week later.
  Other Names: Non-Opioid
  Arms: Non-Opioid Group

SUMMARY:
The purpose of this research study is to compare how well two medications work to control post-operative pain.

DETAILED DESCRIPTION:
This will be a randomized double blinded control trial with subjects randomized to either opioid group (Norco 5-325 milligram) or a non-opioid group (Ibuprofen 400 milligram). Subjects with a renal stones who are consented for a ureteroscopy will be eligible for the study. Subjects eligible for the study will have a discussion with the study team member about treatment options. Subjects can either elect not to be in the study and actively choose which treatment is preferable, or the subject can choose to enter the study and be randomized to one of these treatment arms. The ureteroscopy will be performed using standard of care instruments and techniques. No changes to operative technique will be performed for subjects in the study vs regular patients undergoing the same procedure. Post operatively; investigators plan to discharge all subjects home from the recovery unit. All subjects will be seen one week after surgery for follow up, questioner filling and stent removal.

ELIGIBILITY:
Inclusion Criteria:

* Ureteroscopy performed for renal stones
* Age over 18 years
* Two kidneys

Exclusion Criteria:

* Solitary Kidney
* Poor kidney function (GFR<30)
* Allergy to either Ibuprofen or Norco
* Pelvic Kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gutierrez-Aceves, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We will not share.

REFERENCES:
- [Background] Finney RP. Experience with new double J ureteral catheter stent. J Urol. 1978 Dec;120(6):678-81. doi: 10.1016/s0022-5347(17)57326-7. PMID 731804
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART II. J Urol. 2016 Oct;196(4):1161-9. doi: 10.1016/j.juro.2016.05.091. Epub 2016 May 27. PMID 27238615
- [Background] Joshi HB, Okeke A, Newns N, Keeley FX Jr, Timoney AG. Characterization of urinary symptoms in patients with ureteral stents. Urology. 2002 Apr;59(4):511-6. doi: 10.1016/s0090-4295(01)01644-2. PMID 11927301
- [Background] Mosli HA, Farsi HM, al-Zimaity MF, Saleh TR, al-Zamzami MM. Vesicoureteral reflux in patients with double pigtail stents. J Urol. 1991 Oct;146(4):966-9. doi: 10.1016/s0022-5347(17)37976-4. PMID 1895452
- [Background] Chew BH, Knudsen BE, Nott L, Pautler SE, Razvi H, Amann J, Denstedt JD. Pilot study of ureteral movement in stented patients: first step in understanding dynamic ureteral anatomy to improve stent comfort. J Endourol. 2007 Sep;21(9):1069-75. doi: 10.1089/end.2006.0252. PMID 17941789
- [Background] Al-Kandari AM, Al-Shaiji TF, Shaaban H, Ibrahim HM, Elshebiny YH, Shokeir AA. Effects of proximal and distal ends of double-J ureteral stent position on postprocedural symptoms and quality of life: a randomized clinical trial. J Endourol. 2007 Jul;21(7):698-702. doi: 10.1089/end.2007.9949. PMID 17705753
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846
- [Background] Theisen K, Jacobs B, Macleod L, Davies B. The United States opioid epidemic: a review of the surgeon's contribution to it and health policy initiatives. BJU Int. 2018 Nov;122(5):754-759. doi: 10.1111/bju.14446. Epub 2018 Jul 26. PMID 29896932
- [Background] Large T, Heiman J, Ross A, Anderson B, Krambeck A. Initial Experience with Narcotic-Free Ureteroscopy: A Feasibility Analysis. J Endourol. 2018 Oct;32(10):907-911. doi: 10.1089/end.2018.0459. Epub 2018 Sep 12. PMID 30039709
- [Background] Sobel DW, Cisu T, Barclay T, Pham A, Callas P, Sternberg K. A Retrospective Review Demonstrating the Feasibility of Discharging Patients Without Opioids After Ureteroscopy and Ureteral Stent Placement. J Endourol. 2018 Nov;32(11):1044-1049. doi: 10.1089/end.2018.0539. Epub 2018 Oct 23. PMID 30244594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Group | Non-Opioid Group
Started | 12 | 10
Completed | 7 | 3
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Population: 12 patients were lost to follow up and as such were not included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Group | Non-Opioid Group | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Full Range); unit: years] | 57 [28 to 76] | 53 [39 to 71] | 56 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Amount of Pain Medication Used
Description: Number of tablets taken after surgery
Time Frame: between baseline through day 7
Population: 12 subjects out of total 22 enrolled were lost to follow up
Measure: Mean (Full Range); unit: tablets
Arm/Group | Opioid Group | Non-Opioid Group
Number analyzed (Participants) | 7 | 3
tablets | 7.3 [3 to 25] | 6.67 [0 to 11]

2. Primary Outcome: Number of Subjects Who Need Additional Pain Medication and/or Refill
Description: Number of Subjects Who Need Additional Pain medication and/or Refill
Time Frame: baseline through day 7
Population: 12 subjects out of total 22 enrolled were lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Group | Non-Opioid Group
Number analyzed (Participants) | 7 | 3
Participants | 0 | 0

3. Secondary Outcome: Urinary Index
Description: Ureteral stent symptom questionnaire Urinary Symptom score ranges from 11 to 56 with a higher score denoting a worse outcome.
Time Frame: day 7
Population: 12 subjects out of total 22 enrolled were lost to follow up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Opioid Group | Non-Opioid Group
Number analyzed (Participants) | 7 | 3
score on a scale | 29.2 [20 to 42] | 22.3 [16 to 27]

ADVERSE EVENTS:
Time Frame: baseline through month 6
Arm/Group | Opioid Group | Non-Opioid Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 0/7 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03872843/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT03872843/Prot_SAP_001.pdf